CLINICAL TRIAL: NCT02985866
Title: Clinical Acceptance of the Artificial Pancreas: the International Diabetes Closed Loop (iDCL) Trial: A Randomized Clinical Trial to Assess the Efficacy of Adjunctive Closed Loop Control Versus Sensor-Augmented Pump Therapy in the Management of Type 1 Diabetes
Brief Title: The International Diabetes Closed Loop (iDCL) Trial: Protocol 1
Acronym: iDCL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Jaeb Center for Health Research (Other); TypeZero Technologies (Industry); DexCom, Inc. (Industry); Roche Diagnostic Ltd. (Industry); Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: iDCL; UC4DK108483 (NIH)
Record Dates: First submitted 2016-12-05; First posted 2016-12-07 (Estimated); Results first posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Type1 Diabetes Mellitus
Keywords: Artificial Pancreas; Closed Loop Control; Continuous Glucose Monitor (CGM); inControl Diabetes Management Platform
MeSH Terms: interventions — Pancreas, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Artificial Pancreas (Experimental): Subjects will be provided the Artificial Pancreas (AP) system which includes the inControl Diabetes Management Platform, a study insulin pump, study continuous glucose monitor (CGM), and a study glucometer. This AP system is designed to help control blood sugar in people living with type 1 diabetes.
  Interventions: Device: Artificial Pancreas
- Sensor Augmented Therapy (Active Comparator): Subjects will continue to use their personal insulin pump with a study continuous glucose monitor (CGM) and study glucometer.
  Interventions: Other: Sensor Augmented Therapy

INTERVENTIONS:
Device: Artificial Pancreas — Use of CTR at home for 3 months
  Other Names: Control-to-Range (CTR) closed-loop (CL)
  Arms: Artificial Pancreas
Other: Sensor Augmented Therapy — Use of personal pump with study CGM & glucometer at home for 3 months
  Other Names: SAP
  Arms: Sensor Augmented Therapy

SUMMARY:
The objective of the study is to assess the efficacy and safety of home use of a Control-to-Range (CTR) closed-loop (CL) system.

DETAILED DESCRIPTION:
The protocol is a 3-month parallel group multi-center randomized trial designed to compare Control-to-Range (CTR) closed-loop (CL) with sensor augmented pump therapy (SAP). Approximately 126 subjects will be entered into the randomized trial at approximately seven clinical sites in the United States, such that at least 110 subjects complete the randomized trial. A maximum of 200 subjects may be enrolled in the study in order to achieve the goal of randomizing 126 subjects.

In order to have a broad range of glycemic control among the subjects, a study goal will be to have a minimum of 50 subjects with HbA1c ≥ 7.5% and 50 with HbA1c < 7.5%.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least one year and using insulin for at least 1 year
2. Use of an insulin pump for at least 6 months
3. Age ≥14 years old
4. HbA1c level <10.5% at screening
5. For females, not currently known to be pregnant
6. Willingness not to add glucose-lowering agents (such as Pramlintide, Metformin, GLP-1 analogs, SGLT2 inhibitors) during the study
7. Willingness, if not assigned to the closed-loop group, to avoid use of any closed-loop control system for the duration of the clinical trial
8. Willingness to suspend use of any personal CGM for the duration of the clinical trial once the unblinded study CGM is in use
9. Willingness to establish network connectivity on at least a weekly basis either via local Wifi network or via a study-provided cellular service
10. Currently using no insulins other than one of the following rapid-acting insulins at the time of enrollment: insulin lispro (Humalog), insulin aspart (Novolog), or insulin glulisine (Apidra)
11. Investigator has confidence that the subject can successfully operate all study devices and is capable of adhering to the protocol
12. For subjects less than 18 years old, living with one or more parent/legal guardian (referred to subsequently as diabetes care partner) committed to participating in study training for emergency procedures for severe hypoglycemia and able to contact the subject in case of an emergency

Exclusion Criteria:

1. Medical need for chronic acetaminophen
2. Use of any glucose-lowering agent (such as Pramlintide, Metformin, GLP-1 analogs, SGLT2 inhibitors) in the 3 months prior to enrollment
3. Hemophilia or any other bleeding disorder
4. A condition, which in the opinion of the investigator or designee, would put the participant or study at risk including any contraindication to the use of any of the study devices per FDA labeling
5. Participation in another pharmaceutical or device trial at the time of enrollment or during the study
6. Use of a closed-loop system within the last month prior to enrollment
7. Employed by, or having immediate family members employed by TypeZero Technologies, LLC

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2018-09-04 (Actual); Study Completion 2018-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boris P. Kovatchev, PhD, Principal Investigator — University of Virginia Center for Diabetes Technology; Stacey M. Anderson, MD, Study Chair — University of Virginia Center for Diabetes Technology
Locations (7):
- United States (7):
  - William Sansum Diabetes Center, Santa Barbara, California
  - Stanford University, Stanford, California
  - Barbara Davis Center, University of Colorado, Aurora, Colorado
  - Harvard University (Joslin Diabetes Center), Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Virginia Center for Diabetes Technology, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
NIH's Data Sharing Policy on sharing research resources for research purposes to the scientific community will be followed. Data will be stored in a Data Archive Database includes CGM-insulin delivery time series, meal content, boluses, & exercise will be deidentified & retrievable only by subject ID number. Individual patterns of demographic & insulin treatment parameters leave open a remote possibility of deductive disclosure of subjects with unusual characteristics. Thus, data will be made available only under a Data-Sharing Agreement that includes: (1) a commitment to using the data only for research purposes & not to identify participants; (2) a commitment to securing the data using appropriate computer technology; & (3) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Background] Kovatchev B, Anderson SM, Raghinaru D, Kudva YC, Laffel LM, Levy C, Pinsker JE, Wadwa RP, Buckingham B, Doyle FJ 3rd, Brown SA, Church MM, Dadlani V, Dassau E, Ekhlaspour L, Forlenza GP, Isganaitis E, Lam DW, Lum J, Beck RW; iDCL Study Group. Erratum. Randomized Controlled Trial of Mobile Closed-Loop Control. Diabetes Care 2020;43:607-615. Diabetes Care. 2020 Jun;43(6):1366. doi: 10.2337/dc20-er06. Epub 2020 Apr 3. No abstract available. PMID 32245747
- [Result] Kovatchev B, Anderson SM, Raghinaru D, Kudva YC, Laffel LM, Levy C, Pinsker JE, Wadwa RP, Buckingham B, Doyle FJ 3rd, Brown SA, Church MM, Dadlani V, Dassau E, Ekhlaspour L, Forlenza GP, Isganaitis E, Lam DW, Lum J, Beck RW; iDCL Study Group. Randomized Controlled Trial of Mobile Closed-Loop Control. Diabetes Care. 2020 Mar;43(3):607-615. doi: 10.2337/dc19-1310. Epub 2020 Jan 14. PMID 31937608

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This parallel-group, multicenter, randomized unblinded clinical trial was conducted at 7 US university centers. Participants were diagnosed with type 1 diabetes, treated with insulin for at least 1 year, using pump therapy for at least 6 months, age 14 and above, & HbA1c <10.5% (91 mmol/mol). A study goal was to have at least 50 participants with HbA1c<7.5% (58 mmol/mol) and at least 50 participants with HbA1c >7.5% (58 mmol/mol). Participants were screened October 2017 - May 2018.
Pre-assignment Details: Participants who used a personal Dexcom G4 or G5 CGM pre-study for at least 21 of the prior 28 days proceeded directly to randomization. For these participants, the data downloaded from the personal CGM provided the 2-week baseline data. All others wore a blinded study CGM for 2 weeks to collect baseline data, followed by 2 weeks of training using an unblinded study CGM. Successful completion of the run-in was followed by randomization.
Groups:
- Artificial Pancreas (Closed Loop Control): Subjects will be provided the Artificial Pancreas (AP) system which includes the inControl Diabetes Management Platform, a study insulin pump, study continuous glucose monitor (CGM), and a study glucometer. This AP system is designed to help control blood sugar in people living with type 1 diabetes.
  Artificial Pancreas: Use of CTR at home for 3 months
Period: Overall Study
Arm/Group | Artificial Pancreas (Closed Loop Control) | Sensor Augmented Therapy
Started | 65 | 62
Completed | 64 | 61
Not Completed | 1 | 1
Not completed — Poor CGM data | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Artificial Pancreas (Closed Loop Control) | Sensor Augmented Therapy | Total
Number analyzed (Participants) | 65 | 62 | 127
Age, Customized [Count of Participants; unit: Participants]
  <21 | 18 | 17 | 35
  21 to <35 | 19 | 21 | 40
  35 to <65 | 25 | 21 | 46
  ≥65 | 3 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 28 | 60
  Male | 33 | 34 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 9
  Not Hispanic or Latino | 59 | 59 | 118
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 55 | 55 | 110
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 3 | 0 | 3
Diabetes duration at randomization (years) [Count of Participants; unit: Participants]
  1 to <5 | 10 | 3 | 13
  5 to <10 | 10 | 5 | 15
  10 to <20 | 13 | 29 | 42
  20 to <30 | 18 | 13 | 31
  30 to <40 | 6 | 9 | 15
  ≥40 | 8 | 3 | 11
Prior CGM use [Count of Participants; unit: Participants]
  Never | 1 | 4 | 5
  In past, but not current | 16 | 14 | 30
  Current | 48 | 44 | 92
BMI at enrollment (kg/m2) [Count of Participants; unit: Participants]
  <18 | 2 | 0 | 2
  18 to <25 | 22 | 29 | 51
  25 to <30 | 23 | 22 | 45
  ≥30 | 18 | 11 | 29
HbA1c at randomization: laboratory [Count of Participants; unit: Participants]
  <7.0% (53 mmol/ml) | 22 | 21 | 43
  7.0% to <7.5% (53 to <58 mmol/mol) | 11 | 12 | 23
  7.5% to <8.0% (58 to <64 mmol/mol) | 13 | 15 | 28
  8.0% to ≤10.5% (64 to ≤91 mmol/mol) | 19 | 14 | 33
C-Peptide at randomization (nmol/L): Laboratory [Count of Participants; unit: Participants]
  <0.003 | 48 | 45 | 93
  0.003 to <0.1 | 9 | 13 | 22
  0.1 to <0.5 | 6 | 4 | 10
  ≥0.5 | 2 | 0 | 2
Diabetes ketoacidosis events in the last 12 months [Count of Participants; unit: Participants]
  0 | 64 | 61 | 125
  1 | 1 | 0 | 1
  2 | 0 | 1 | 1
Severe hypoglycemic events in past 12 months [Count of Participants; unit: Participants]
  0 | 63 | 58 | 121
  1 | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Time Below 70 mg/dL
Description: CGM-measured % time below 70 mg/dL - 1st co-primary outcome (superiority)
Time Frame: Post randomization (final 11 weeks)
Measure: Mean (Standard Deviation); unit: percentage of total CGM time
Arm/Group | Artificial Pancreas (Closed Loop Control) | Sensor Augmented Therapy
Number analyzed (Participants) | 64 | 61
percentage of total CGM time | 2.4 (1.7) | 4.0 (3.4)
Statistical Analysis 1: Comparison: Artificial Pancreas (Closed Loop Control) vs Sensor Augmented Therapy; Statistical analyses were performed on an intention-to-treat basis, and all participants with any amount of post randomization data were included in all analyses; Test type: Superiority — The first co-primary end point was superiority of CLC over SAP in terms of CGM-measured time below 70 mg/dL. The treatment groups were compared using linear models while adjusting for age, corresponding baseline value, previous CGM use, and a random center effect. Missing baseline data were handled by direct likelihood method. Model residuals were confirmed to be approximately normally distributed; p < 0.0001, Mixed Models Analysis — To address the issue of multiple comparisons with 2 primary outcomes, the intervention was considered effective only if both co-primary outcomes were statistically significant at 5% level. P value for noninferiority NI (prespecified NI limit = 5%); The groups were compared using linear models while adjusting for age, corresponding baseline value, previous CGM use, and a random center effect

2. Primary Outcome: Time Above 180 mg/dL
Description: CGM-measured % time above 180 mg/dL - 2nd co-primary outcome (noninferiority)
Time Frame: Post randomization (final 11 weeks)
Measure: Mean (Standard Deviation); unit: percentage of total CGM time
Arm/Group | Artificial Pancreas (Closed Loop Control) | Sensor Augmented Therapy
Number analyzed (Participants) | 64 | 61
percentage of total CGM time | 34 (11) | 39 (15)
Statistical Analysis 1: Comparison: Artificial Pancreas (Closed Loop Control) vs Sensor Augmented Therapy; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — The second co-primary end point was noninferiority in CGM-measured time above 180 mg/dL, with a noninferiority limit of 5%. The treatment groups were compared using linear models while adjusting for age, corresponding baseline value, previous CGM use, and a random center effect. Missing baseline data were handled by direct likelihood method. Model residuals were confirmed to be approximately normally distributed; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Time Below 54 mg/dL
Description: Percent time CGM readings were below 54 mg/dL
Time Frame: Post randomization (final 11 weeks)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Artificial Pancreas | Sensor Augmented Therapy
Number analyzed (Participants) | 64 | 61
Percentage | 0.6 (0.6) | 1.1 (1.2)
Statistical Analysis 1: Comparison: Artificial Pancreas vs Sensor Augmented Therapy; Same as for the primary outcomes; Test type: Superiority — Same as for primary outcome 1; p < 0.05, Mixed Models Analysis — All secondary analyses were corrected for multiple comparisons using the false discovery rate at a 10% level for statistical significance. All secondary P values reported are two-sided; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Time Below 60 mg/dL
Description: CGM-measured % time below 60 mg/dL
Time Frame: Post randomization (final 11 weeks)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Artificial Pancreas (Closed Loop Control) | Sensor Augmented Therapy
Number analyzed (Participants) | 64 | 61
Percentage | 1.1 (1.0) | 1.9 (1.9)
Statistical Analysis 1: Comparison: Artificial Pancreas (Closed Loop Control) vs Sensor Augmented Therapy; Same as for the primary outcomes; Test type: Superiority — Same as for primary outcome 1; p < 0.05, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]

5. Secondary Outcome: Time in Range 70-180 mg/dL
Description: CGM-measured % in range 70-180 mg/dL
Time Frame: Post randomization (final 11 weeks)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Artificial Pancreas (Closed Loop Control) | Sensor Augmented Therapy
Number analyzed (Participants) | 64 | 61
Percentage | 64 (11) | 57 (14)
Statistical Analysis 1: Comparison: Artificial Pancreas (Closed Loop Control) vs Sensor Augmented Therapy; Same as for the primary outcomes; Test type: Superiority — Same as for primary outcome 1; p < 0.05, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]

6. Secondary Outcome: Time in Range 70-140 mg/dL
Description: CGM-measured % time in range 70-140 mg/dL
Time Frame: Post randomization (final 11 weeks)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Artificial Pancreas (Closed Loop Control) | Sensor Augmented Therapy
Number analyzed (Participants) | 64 | 61
Percentage | 39 (10) | 35 (12)
Statistical Analysis 1: Comparison: Artificial Pancreas (Closed Loop Control) vs Sensor Augmented Therapy; Same as for the primary outcomes; Test type: Superiority — Same as for primary outcome 1; p < 0.05, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]

7. Secondary Outcome: Time Above 250 mg/dL
Description: CGM-measured % time above 250 mg/dL
Time Frame: Post randomization (final 11 weeks)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Artificial Pancreas (Closed Loop Control) | Sensor Augmented Therapy
Number analyzed (Participants) | 64 | 61
Percentage | 11.2 (7.4) | 13.7 (11.4)
Statistical Analysis 1: Comparison: Artificial Pancreas (Closed Loop Control) vs Sensor Augmented Therapy; Same as for the primary outcomes; Test type: Superiority — Same as for primary outcome 1; p < 0.05, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]

8. Secondary Outcome: Time Above 300 mg/dL
Description: CGM-measured % time above 300 mg/dL
Time Frame: Post randomization (final 11 weeks)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Artificial Pancreas (Closed Loop Control) | Sensor Augmented Therapy
Number analyzed (Participants) | 64 | 61
Percentage | 4.4 (4.2) | 5.7 (7.1)
Statistical Analysis 1: Comparison: Artificial Pancreas (Closed Loop Control) vs Sensor Augmented Therapy; Same as for the primary outcomes; Test type: Superiority — Same as for primary outcome 1; p < 0.05, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]

9. Secondary Outcome: Coefficient of Variation
Description: CGM-measured coefficient of variation (CV)
Time Frame: Post randomization (final 11 weeks)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Artificial Pancreas (Closed Loop Control) | Sensor Augmented Therapy
Number analyzed (Participants) | 64 | 61
Percentage | 37 (5) | 38 (5)
Statistical Analysis 1: Comparison: Artificial Pancreas (Closed Loop Control) vs Sensor Augmented Therapy; Same as for the primary outcomes; Test type: Superiority — Same as for primary outcome 1; p < 0.05, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 13 weeks
Arm/Group | Artificial Pancreas (Closed Loop Control) | Sensor Augmented Therapy
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/62
Serious Adverse Events (participants affected / at risk) | 1/65 | 0/62
Other Adverse Events (participants affected / at risk) | 0/65 | 2/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Artificial Pancreas (Closed Loop Control) (N=65) | Sensor Augmented Therapy (N=62)
Hypoglycemic seizure (Nervous system disorders) | 1 (1) | 0 (0) — Severe hypoglycemia on 2/26/18 at ~5:30PM. Spouse noticed convulsion during sleep CGM reading = 50 mg/dl. Spouse provided two boxes of juice & glucose tablets. Participant doesn't recall episode. Complete recovery after rescue carbohydrates.
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Participant ran 100k race on 5/12/18.Felt overheated & vomiting x2 after 52.8 miles (13.5h run time). Admitted to the ER for dehydration & DKA risk. BG in 200s & ketones were negative. Complete recovery.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Artificial Pancreas (Closed Loop Control) (N=65) | Sensor Augmented Therapy (N=62)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) — Nausea & vomiting started 02/13/18. No fever. Exposed GI illness day before. Blood glucose=99 mg/dl; serum ketones=1.2 mmol/L. In follow up call, ketones=1.1 mmol/L one hour later. On 02/14/18, ketones=0.3 mmol/L. Complete recovery.
Surgery (Surgical and medical procedures) | 0 (0) | 1 (1) — Planned in-patient surgery on 4/10/18. Removal of Whartin growth behind left ear. Complete recovery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/66/NCT02985866/Prot_SAP_002.pdf
  • Informed Consent Form (2018-04-06): https://cdn.clinicaltrials.gov/large-docs/66/NCT02985866/ICF_001.pdf